CLINICAL TRIAL: NCT01179399
Title: A Phase 1, Open-Label, Dose-Escalation Study of Orally Administered TAK-960, a Polo-Like Kinase 1 Inhibitor, in Patients With Advanced Nonhematologic Malignancies
Brief Title: Study of Orally Administered TAK-960 in Patients With Advanced Nonhematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C22001
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Nonhematological Malignancies
MeSH Terms: interventions — 4-((9-cyclopentyl-7,7-difluoro-5-methyl-6-oxo-6,7,8,9-tetrahydro-5H-pyrimido(4,5-b)(1,4)diazepin-2-yl)amino)-2-fluoro-5-methoxy-N-(1-methylpiperidin-4-yl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-960 (Experimental)
  Interventions: Drug: TAK-960

INTERVENTIONS:
Drug: TAK-960 — TAK-960 administered orally once a day for 21-days of a 28-day treatment cycle. A 3 + 3 dose escalation scheme will be employed.

SUMMARY:
Overview of Study Design: This is a phase 1, multicenter, open-label, multiple-dose, dose-escalation study designed to evaluate the safety, tolerability, pharmacokinetics (PK), and antitumor activity of TAK-960 in patients with advanced nonhematologic malignancies. This study will be the first to administer TAK-960 to humans. The patient population will consist of adults with a nonhematologic malignancy for which standard treatment is no longer effective or does not offer curative or life-prolonging potential, or for which no standard treatment is available.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Male or female 18 years or older
* Clinical laboratory values as specified in protocol
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically and/or cytologically confirmed diagnosis of metastatic, unresectable, advanced evaluable nonhematologic malignancy for which standard treatment is not available or no longer effective
* Radiographically or clinically evaluable tumor
* Suitable venous access for study-required blood sampling
* Female patients who are postmenopausal, surgically sterile or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse
* Male patients who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse
* Voluntary written consent
* Willing to undergo biopsy procedures (expansion phase only)
* Weight at least 40 kg
* Recovered from the reversible effects of prior antineoplastic therapy to Grade ≤ 1 or to patient's baseline values, excluding alopecia

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Diagnosis of primary central nervous system malignancy or carcinomatous meningitis
* Patient has symptomatic brain metastasis. Patients with brain metastases must: have stable neurologic status for at least 2 weeks following completion of local therapy AND be without neurologic dysfunction that would confound the evaluation of adverse events
* Prior allogeneic bone marrow or stem cell transplant
* Prior therapy or treatment as specified in protocol
* Female patients who are lactating or who have a positive serum pregnancy test during the screening period of within 3 days before the first dose of TAK-960
* Myocardial infarction within 6 months before first dose of TAK-960
* Any of the cardiovascular conditions or values as specified in the study protocol within 6 months before the first dose of TAK-960
* Infection requiring systemic anti-infective therapy within 14 days before the start of TAK-960, or other severe infection
* Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive or known suspected active hepatitis C infection
* A diagnosis of or treated for another malignancy within 2 years before the first dose of TAK-960 or previous diagnosis of another malignancy and any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Any serious medical or psychiatric illness that could potentially interfere with the completion of treatment
* Recurrent nausea or vomiting or requirement for antiemetic therapy within 14 days before the first dose of TAK-960
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerability of TAK-960, including difficulty swallowing capsules
* Treatment with any investigational products within 21 days before the first dose of TAK-960
* Systemic use of strong CYP3A inhibitors or inducers within 14 days before the first dose of TAK-960
* Patients enrolled in the expansion cohorts where tumor biopsies are required must meet additional criteria according to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- TAK-960: Given orally (PO) for 21 days of a 28-day treatment cycle.
Period: Overall Study
Arm/Group | TAK-960
Started | 32
Completed | 0
Not Completed | 32
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 30
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | TAK-960
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 20
  Spain | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of TAK-960
Description: Adverse events, serious adverse events, assessments of clinical laboratory values, vital sign measurements and electrocardiograms (ECGs)
Time Frame: up to 12 months
Population: Maximum tolerable dose (MTD) and recommended phase 2 dose (RP2D) of TAK-960 were not determined due to sponsor decision to discontinue the study for business reasons.
Arm/Group | TAK-960
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | TAK-960
Serious Adverse Events (participants affected / at risk) | 13/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-960 (N=32)
Anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Device related infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-960 (N=32)
Nausea (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 5
Gamma-glutamyltransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pyrexia (General disorders) | 3
Oedema peripheral (General disorders) | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pollakiuria (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No